CLINICAL TRIAL: NCT02978040
Title: Facilitation Through Aggrastat or Cangrelor Bolus and Infusion Over prasugreL: a mUlticenter Randomized Open-label Trial in patientS With ST-elevation Myocardial inFarction Referred for primAry percutaneouS inTERvention.FABOLUS FASTER Trial
Brief Title: Randomized Comparison of Cangrelor, Tirofiban and Prasugrel in Patients With STEMI Referred for Primary PCI.
Acronym: FABOLUS-FASTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FABOLUS-FASTER
Record Dates: First submitted 2016-11-17; First posted 2016-11-30 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease; STEMI - ST Elevation Myocardial Infarction
Keywords: Antiplatelet therapy; Cangrelor; Tirofiban; Prasugrel; Acute Myocardial Infarction; Primary Percutaneous Coronary Intervention; Pharmacokinetic/Pharmacodynamic
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction | interventions — cangrelor; Tirofiban; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study is open label. Participant and Investigators will be not masked to randomly assigned treatments. An independent blinded committee will assess clinical adverse events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cangrelor (Experimental): Cangrelor bolus of 30 µg/Kg followed by infusion at 4 µg/Kg/min for 2 h (or to the end of PCI).
  Interventions: Drug: Cangrelor
- Tirofiban (Active Comparator): Tirofiban bolus of 25 µg/Kg bolus followed by infusion at 0.15 µg/Kg/min for 2 h (or to the end of PCI) (infusion rate of 0.075 µg/Kg/min for patients with creatinine clearance < 60 ml/min).
  Interventions: Drug: Tirofiban
- Prasugrel (Active Comparator): Prasugrel oral integer or chewed at an identical loading dose of 60 mg
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Cangrelor — Cangrelor will be administered as bolus of 30 µg/Kg followed by infusion at 4 µg/Kg/min for 2 h (or to the end of PCI); at the end of infusion, oral prasugrel at loading dose of 60 mg will be administrated, then 10 mg daily (5 mg daily if body weight < 60 kg or age > 75 years old).
  Other Names: Kengreal; Kengrexal
  Arms: Cangrelor
Drug: Tirofiban — Tirofiban will be administrated as 25 µg/Kg bolus followed by infusion at 0.15 µg/Kg/min for 2 h (or to the end of PCI) (infusion rate of 0.075 µg/Kg/min for patients with creatinine clearance < 60 ml/min); at the end of infusion, oral prasugrel at loading dose of 60 mg will be administrated, then 10 mg daily (5 mg daily if body weight < 60 kg or age > 75 years old) .
  Other Names: Aggrastat
  Arms: Tirofiban
Drug: Prasugrel — In the prasugrel arm no intravenous anti-platelet drug will be administered. Patients will be randomized to oral integer prasugrel or chewed oral prasugrel at an identical loading dose of 60 mg, then 10 mg daily (5 mg daily if body weight < 60 kg or age > 75 years old).
  Other Names: Efient
  Arms: Prasugrel

SUMMARY:
Primary percutaneous coronary intervention (PCI) is the main reperfusion therapy in patients with ST-elevation myocardial infarction (STEMI). The optimal platelet inhibition at the time of PCI is fundamental, however, the comparative speed of action of cangrelor as opposed to tirofiban and to chewed or integer loading dose of prasugrel is unknown.

The purpose of this trial is to assess the inhibition of platelet aggregation with different regimens on platelet inhibition (tirofiban bolus+infusion, cangrelor bolus+infusion, prasugrel chewed loading dose, prasugrel integer loading dose) in the early phase of primary PCI.

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention (PCI) is the main reperfusion therapy in patients with ST-elevation myocardial infarction (STEMI). Ancillary pharmacological therapy includes dual antiplatelet therapy with aspirin and an inhibitor of P2Y12 receptor, responsible of adenosine diphosphate(ADP)-mediated platelet activation.Prasugrel and ticagrelor are the most recent and efficient oral P2Y12 inhibitors available to date. However, in STEMI even prasugrel and ticagrelor could have a significant delay of onset of action. Early in-ambulance administration can increase the inhibition of P2Y12 receptor, however, the benefits versus risks balance remain uncertain. Recently, small-scale independent studies suggested that chewed or crushed loading dose of ticagrelor or prasugrel can achieve more pronounced platelet inhibition compared with standard whole tablets soon after drug administration. Yet, the delay in platelet inhibition remains considerable even after chewed or crushed loading dose of newer oral P2Y12 inhibitors and suboptimal modulation of platelet reactivity at the time of primary intervention may persist. Tirofiban and cangrelor are intravenous drugs with a more rapid onset and offset of action compared with oral agents. Both agents have been extensively tested in clinical trials including patients with STEMI. However, the comparative speed of action of cangrelor as opposed to tirofiban and to chewed or integer loading dose of prasugrel is unknown. The proposed investigation will have a prospective, randomized, design in which STEMI patients undergoing primary PCI will be randomized to receive Cangrelor or Tirofiban or Prasugrel (these patients will be further randomized to receive chewed or integer tablets). Pharmacodynamic testing will be performed at several time points to test the investigators' study hypotheses: 1) Cangrelor will have similar inhibitory effect to Tirofiban (non-inferiority of Cangrelor compared with Tirofiban); 2) Compared with Prasugrel, Cangrelor and Tirofiban will achieve more prompt and enhanced platelet inhibitory effects (superiority of both Tirofiban and Cangrelor to integer Prasugrel); 3) Compared with integer loading dose of Prasugrel, chewed Prasugrel regimen will achieve more prompt and enhanced platelet inhibitory effects (superiority of chewed Prasugrel to integer Prasugrel). This study will provide insights on the pharmacodynamic effects of these drugs and will help clinicians choose the most appropriate treatment to avoid complications related to inadequate platelet inhibition in the early phase of patients with STEMI undergoing primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* ST-segment elevation myocardial infarction
* Referred for primary PCI either within 12 h of symptom onset or between 12 and 24 h after onset with evidence of continuing ischemia

Exclusion Criteria:

* Unconsciousness
* Other conditions that make the patient incapable receiving integer loading dose of prasugrel
* Any contraindication and/or known hypersensitivity or allergy to aspirin, prasugrel, intravenous unfractionated heparin, cangrelor, tirofiban
* Any contraindication to primary PCI
* Administration of glycoprotein IIb/IIIa inhibitors (GPI) or P2Y12-inhibitors or cangrelor < 7 days
* Chronic dialysis
* Recent (< 15 days) or current major bleeding
* Recent (< 15 days) major surgery
* Administration of fibrinolytics < 30 days
* Current use or indication to oral anticoagulant
* Previous stroke or transient ischemic attack (TIA)
* Inability to follow the procedures of the study (language problems, psychological disorders, dementia) or comorbidities associated with less than 6 months survival (active malignancies drug or alcohol abuse, etc.)
* Women who are pregnant or breast feeding or with potential to become pregnant during the course of the study (age < 55 years and last menstruation within the last 12 months) and did not undergo tubal ligation, ovariectomy or hysterectomy
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Inhibition of platelet activity (IPA, %) with LTA-ADP 20 µmol/l | 30 minutes
  Primary outcome is platelet inhibition assessed with light transmission aggregometry (LTA) in platelet rich plasma with the addition of adenosine diphosphate (ADP) 20 µmol/l at 30 minutes from drug administration

SECONDARY OUTCOMES:
Inhibition of platelet activity (IPA, %) with LTA-ADP 20 µmol/l | 15 minutes, 1 hour, 2 hours, 3 hours, 4-6 hours
  Platelet inhibition assessed with light transmission aggregometry (LTA) in platelet rich plasma with the addition of ADP 20 µmol/l at 15 minutes, 1h, 2h, 3h and 4-6h from drug administration
Inhibition of platelet activity (IPA, %) with LTA-ADP 5 µmol/l | 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4-6 hours
  Platelet inhibition assessed with light transmission aggregometry (LTA) in platelet rich plasma with the addition of ADP 5 µmol/l at 15 minutes, 30 minutes, 1h, 2h, 3h and 4-6h from drug administration
Inhibition of platelet activity (IPA, %) with LTA-TRAP 5 µmol/l | 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4-6 hours
  Platelet inhibition assessed with light transmission aggregometry (LTA) in platelet rich plasma with the addition of thrombin receptor-activating peptides (TRAP) 5 µmol/l at 15 minutes, 30 minutes, 1h, 2h, 3h and 4-6h from drug administration
Inhibition of platelet activity (IPA, %) with LTA-TRAP 15 µmol/l | 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4-6 hours
  Platelet inhibition assessed with light transmission aggregometry (LTA) in platelet rich plasma with the addition of TRAP 15 µmol/l at 15 minutes, 30 minutes, 1h, 2h, 3h and 4-6h from drug administration
Area under the curve (AUC) at Multiplate with ADP test | 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4-6 hours
  Platelet inhibition assessed with Multiplate ADP test at 15 minutes, 30 minutes, 1h, 2h, 3h and 4-6h from drug administration
Area under the curve (AUC) at Multiplate with TRAP test | 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4-6 hours
  Platelet inhibition assessed with Multiplate TRAP test at 15 minutes, 30 minutes, 1h, 2h, 3h and 4-6h from drug administration
Angiographic result | immediately after PCI procedure
  Final angiographic result evaluated by proportion of patients with TIMI flow<3
Electrocardiographic result | immediately after PCI procedure and 90 minutes after PCI
  ST resolution at ECG recorded after PCI
Infarct size at Cardiac Magnetic Resonance Imaging (MRI) | 3 days and 4-6 months after PCI
  Infarct size assessed at cardiac MRI
Intramyocardial haemorrhage at Cardiac Magnetic Resonance Imaging (MRI) | 3 days and 4-6 months after PCI
  Intramyocardial haemorrhage assessed at cardiac MRI
Major adverse ischemic clinical events | 48 h and 30 days after PCI
  Major adverse ischemic clinical events (including death, cardiac death, myocardial infarction, stroke, urgent target vessel revascularization, definite/probable stent thrombosis and their combinations in composite endpoints) will be evaluated 48 hours and 30 days from primary PCI.
Bleeding events | 48 h and 30 days after PCI
  Bleeding events according to Bleeding Academic Research Consortium (BARC), Thrombolysis in Myocardial Infarction (TIMI), Global Use of Strategies To Open occluded arteries (GUSTO) bleeding scales as well as Net adverse clinical events (NACE; defined as the composite of death, non-fatal myocardial infarction, definite/probable stent thrombosis, non-fatal stroke, and BARC 2, 3, or 5 bleeding) will be evaluated at 48 hours and 30 days from primary PCI

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, Prof, Study Chair — Department of Cardiology, Bern University Hospital; Giuseppe Gargiulo, MD, Principal Investigator — Department of Cardiology, Bern University Hospital
Locations (3):
- Italy (2):
  - University of Ferrara, Ferrara
  - University of Naples Federico II, Naples
- Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Minuz P, Giorgetti A, Meneguzzi A, Taus F, Ribeiro RP, Baldessari F, Gargiulo G, Gragnano F, Landi A, Castelli M, Gottardo R, Bortolotti F, Verlato G, Fava C, Cattaneo M, Tagliaro F, Valgimigli M. Prasugrel Intermediate Metabolite Modulates Platelet Inhibition by Negatively Interfering With an Active Metabolite: An Ex Vivo, In Vitro, and In Silico Study. Arterioscler Thromb Vasc Biol. 2025 May;45(5):792-804. doi: 10.1161/ATVBAHA.124.321916. Epub 2025 Mar 20. PMID 40109258
- [Derived] Gargiulo G, Esposito G, Avvedimento M, Nagler M, Minuz P, Campo G, Gragnano F, Manavifar N, Piccolo R, Tebaldi M, Cirillo P, Hunziker L, Vranckx P, Leonardi S, Heg D, Windecker S, Valgimigli M. Cangrelor, Tirofiban, and Chewed or Standard Prasugrel Regimens in Patients With ST-Segment-Elevation Myocardial Infarction: Primary Results of the FABOLUS-FASTER Trial. Circulation. 2020 Aug 4;142(5):441-454. doi: 10.1161/CIRCULATIONAHA.120.046928. Epub 2020 Jun 27. PMID 32795098
- [Derived] Gargiulo G, Esposito G, Cirillo P, Nagler M, Minuz P, Campo G, Gragnano F, Manavifar N, Piccolo R, Avvedimento M, Tebaldi M, Wahl A, Hunziker L, Billinger M, Heg D, Windecker S, Valgimigli M. Facilitation Through Aggrastat or Cangrelor Bolus and Infusion Over PrasugreL: a MUlticenter Randomized Open-label Trial in PatientS with ST-elevation Myocardial InFarction Referred for PrimAry PercutaneouS InTERvention (FABOLUS FASTER) Trial: Design and Rationale : The FABOLUS FASTER Trial. J Cardiovasc Transl Res. 2021 Feb;14(1):110-119. doi: 10.1007/s12265-020-09969-4. Epub 2020 Feb 24. PMID 32096064